CLINICAL TRIAL: NCT01977794
Title: A Randomized, Comparative Trial of Concor AM, a Fixed Dose Combination of Bisoprolol and Amlodipine, on the Treatment of Essential Hypertensive Patients Whose Blood Pressure is Not Well Controlled by Monotherapy of Bisoprolol 5mg or Amlodipine 5mg
Brief Title: Fixed Dose Combination of Bisoprolol and Amlodipine in the Treatment of Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200006-524
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Bisoprolol; Amlodipine; Fixed dose combination (FDC); Systolic Blood Pressure (SBP); Diastolic Blood Pressure (DBP)
MeSH Terms: conditions — Hypertension | interventions — Bisoprolol; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bisoprolol failed group (Experimental): Subjects who failed monotherapy with bisoprolol 5 milligram (mg) before trial inclusion will be randomized to bisoprolol failed group to receive Bisoprolol/Amlodipine FDC tablet
  Interventions: Drug: Bisoprolol/Amlodipine (Bisoprolol failed group)
- Amlodipine failed group (Experimental): Subjects who failed monotherapy with amlodipine 5 mg before trial inclusion will be randomized to amlodipine failed group to receive Bisoprolol/Amlodipine FDC tablet.
  Interventions: Drug: Bisoprolol/Amlodipine (Amlodipine failed group)

INTERVENTIONS:
Drug: Bisoprolol/Amlodipine (Bisoprolol failed group) — Bisoprolol/Amlodipine FDC tablet will be orally administered at an initial dose of 5 mg/5 mg once daily for 6 weeks. If blood pressure (BP) is controlled at Week 6 (Day 43), the same dose will continue for next 6 weeks. If the BP is not controlled at Day 43, the dose will be increased to Bisoprolol/Amlodipine 5mg/10mg or 10mg/5mg for next 6 weeks. Subjects who have controlled BP at Week 12 (Day 85), will continue with the same dose for next 6 weeks. If their BP is not controlled at Day 85, dose will be increased to the next level (Bisoprolol/Amlodipine 5mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/5mg dose and Bisoprolol/Amlodipine and 10mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/10mg dose) until Week 18 (Day 127).
  Other Names: Concor AM
  Arms: Bisoprolol failed group
Drug: Bisoprolol/Amlodipine (Amlodipine failed group) — Bisoprolol/Amlodipine FDC tablet will be orally administered at an initial dose of 5 milligram (mg)/5 mg once daily for 6 weeks. If BP is controlled at Week 6 (Day 43), the same dose will continue for next 6 weeks. If the BP is not controlled at Day 43, the dose will be increased to Bisoprolol/Amlodipine 5mg/10mg or 10mg/5mg for next 6 weeks. Subjects who have controlled BP at Week 12 (Day 85), will continue with the same dose for next 6 weeks. If their BP is not controlled at Day 85, dose will be increased to the next level (Bisoprolol/Amlodipine 5mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/5mg dose and Bisoprolol/Amlodipine and 10mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/10mg dose) until Week 18 (Day 127).
  Other Names: Concor AM
  Arms: Amlodipine failed group

SUMMARY:
This is a randomized, comparative Phase 3 trial to investigate the efficacy of fixed dose combination (FDC) of bisoprolol and amlodipine in hypertensive subjects (superiority of FDC over monotherapies).

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension not controlled at 5 mg bisoprolol or 5 mg amlodipine at least 4 weeks (definition of not controlled: SBP greater than or equal to (>=) 140 millimeter of mercury (mmHg) with or without DBP >= 90 mmHg)
* Male or female subjects >=18 years of age, without limitation on race
* Medically accepted effective contraception if procreative potential exists (applicable for both male and female subjects until at least 90 days after the last dose of trial treatment)
* Subjects who have signed the informed consent form before any trial related assessment

Exclusion Criteria:

* General contraindications of beta-blockers and/or calcium channel blockers

  * Previous and concurrent acute heart failure or during episodes of heart failure decompensation requiring intravenous inotropic therapy
  * Concurrent cardiogenic shock
  * Previous and concurrent second or third degree atrioventricular (AV) block (without a pacemaker)
  * Previous and concurrent sick sinus syndrome
  * Previous and concurrent sinoatrial block
  * Concurrent symptomatic bradycardia
  * Concurrent symptomatic hypotension
  * Previous and concurrent severe bronchial asthma or chronic obstructive pulmonary diseases
  * Previous and concurrent severe peripheral arterial occlusive diseases and Raynaud's syndrome
  * Untreated pheochromocytoma
  * Concurrent metabolic acidosis
  * Known hypersensitivity to bisoprolol, amlodipine, dihydropyridine derivates or to any of the excipients
* Seated pulse rate less than 60 beats per minute (bpm) at screening
* Any other anti-hypertensive drugs (other than bisoprolol and amlodipine) are used within 4 weeks prior to the screening visit
* Use of any enzyme-modifying drugs acting on cytochrome P450 (CYP) 3A4 enzymes via inhibition (such as ketoconazole, itraconazole, ritonavir) or induction (such as rifampicin or hypericum perforatum) within 28 days before Day 1 of the trial
* Other significant disease that in the Investigator's opinion that would exclude the subject from the trial, such as uncontrolled diabetes mellitus, severe liver and/or kidney dysfunction, decompensated cardiac failure
* Any other condition or therapy which in the Investigator's opinion would pose a risk to the subject or interfere with the trial objectives
* Concurrent alcohol and/or drug abuse
* Known hypersensitivity to the trial treatments
* Pregnancy and lactation period. All female subjects with reproductive potential must have a negative pregnancy serum test within the 7 days prior to enrollment
* Known lack of subject compliance
* Legal incapacity or limited legal capacity
* Participation in another clinical trial within the previous 30 days
* Persons directly involved in the execution of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center located in, Darmstadt, Germany

REFERENCES:
- [Derived] Gottwald-Hostalek U, Li L, Montenegro P. Bisoprolol/amlodipine combination therapy improves blood pressure control in patients with essential hypertension following monotherapy failure. Curr Med Res Opin. 2016 Oct;32(10):1735-1743. doi: 10.1080/03007995.2016.1205573. Epub 2016 Jul 4. PMID 27334671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 clinical trial sites in Guatemala.
Pre-assignment Details: A total of 200 subjects (100 subjects in the amlodipine failed group, and 100 subjects in the bisoprolol failed group) were enrolled and randomized in the trial. Out of which 196 subjects (97 subjects in amlodipine failed group and 99 subjects in bisoprolol failed group) were included in modified intent-to-treat (MITT) analysis set.
Groups:
- Amlodipine Failed Group: Subjects who failed monotherapy with amlodipine 5 milligram (mg) before trial inclusion were randomized to amlodipine failed group to receive Bisoprolol/Amlodipine fixed dose combination(FDC) tablet. Bisoprolol/Amlodipine FDC tablet was orally administered at initial dose of 5mg/5mg once daily for 6 weeks.If blood pressure (BP) was controlled at Week 6(Day 43),same dose continued for next 6 weeks. If BP was not controlled at Day 43,dose was increased to Bisoprolol/Amlodipine 5mg/10mg or 10mg/5mg for next 6 weeks.Subjects who had controlled BP atWeek 12(Day 85),continued same dose that they were receiving for next 6 weeks. If BP was not controlled at Day 85,dose was increased to next level,(Bisoprolol/Amlodipine 5mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/5mg dose and Bisoprolol/Amlodipine 10mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/10mg dose) until Week 18(Day 127).Controlled BP=Systolic BP(SBP)<140 millimetre of mercury(mmHg) and Diastolic BP(DBP)<90mmHg.
- Bisoprolol Failed Group: Subjects who failed monotherapy with bisoprolol 5 mg before trial inclusion were randomized to bisoprolol failed group to receive Bisoprolol/Amlodipine FDC tablet. Bisoprolol/Amlodipine FDC tablet was orally administered at an initial dose of 5 mg/5 mg once daily for 6 weeks. If BP was controlled at Week 6 (Day 43), the same dose was continued for next 6 weeks. If the BP was not controlled at Day 43, the dose was increased to Bisoprolol/Amlodipine 5mg/10mg or 10mg/5mg for next 6 weeks. Subjects who had controlled BP at Week 12 (Day 85), continued with the same dose that they were receiving for next 6 weeks. If their BP was not controlled at Day 85, dose was increased to the next level (Bisoprolol/Amlodipine 5mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/5mg dose and Bisoprolol/Amlodipine and 10mg/10mg for subjects receiving Bisoprolol/Amlodipine 5mg/10mg dose) until Week 18 (Day 127). Controlled BP = SBP <140 mmHg and DBP <90 mmHg.
Period: Overall Study
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group
Started | 100 | 100
Completed | 92 | 94
Not Completed | 8 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 1 | 1
Not completed — Withdrew consent | 2 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: MITT analysis set was defined as all randomized and treated subjects with at least 1 SBP measurement after the date of first dose of investigational medicinal product (IMP).
Groups:
- Amlodipine Failed Group: Subjects who failed monotherapy with amlodipine 5 mg before trial inclusion were randomized to amlodipine failed group to receive Bisoprolol/Amlodipine FDC tablet. Bisoprolol/Amlodipine FDC tablet was orally administered at an initial dose of 5 mg/5 mg once daily for 6 weeks. If BP was controlled at Week 6 (Day 43), the same dose was continued for next 6 weeks. If the BP was not controlled at Day 43, the dose was increased to Bisoprolol/Amlodipine 5 mg/10 mg or 10 mg/5 mg for next 6 weeks. Subjects who had controlled BP at Week 12 (Day 85), continued with the same dose that they were receiving for next 6 weeks. If their BP was not controlled at Day 85, dose was increased to the next level (Bisoprolol/Amlodipine 5 mg/10 mg for subjects receiving Bisoprolol/Amlodipine 5 mg/5 mg dose and Bisoprolol/Amlodipine and 10 mg/10 mg for subjects receiving Bisoprolol/Amlodipine 5 mg/10 mg dose) until Week 18 (Day 127). Controlled BP= SBP <140 mmHg and DBP <90 mmHg.
- Bisoprolol Failed Group: Subjects who failed monotherapy with bisoprolol 5 mg before trial inclusion were randomized to bisoprolol failed group to receive Bisoprolol/Amlodipine FDC tablet. Bisoprolol/Amlodipine FDC tablet was orally administered at an initial dose of 5 mg/5 mg once daily for 6 weeks. If BP was controlled at Week 6 (Day 43), the same dose was continued for next 6 weeks. If the BP was not controlled at Day 43, the dose was increased to Bisoprolol/Amlodipine 5 mg/10 mg or 10 mg/5 mg for next 6 weeks. Subjects who had controlled BP at Week 12 (Day 85), continued with the same dose that they were receiving for next 6 weeks. If their BP was not controlled at Day 85, dose was increased to the next level (Bisoprolol/Amlodipine 5 mg/10 mg for subjects receiving Bisoprolol/Amlodipine 5 mg/5 mg dose and Bisoprolol/Amlodipine and 10 mg/10 mg for subjects receiving Bisoprolol/Amlodipine 5mg/10mg dose) until Week 18 (Day 127). Controlled BP= SBP <140 mmHg and DBP <90 mmHg.
- Total: Total of all reporting groups
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group | Total
Number analyzed (Participants) | 97 | 99 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.62) | 59.6 (12.05) | 61.5 (11.96)
Gender [Count of Participants; unit: Participants]
  Female | 77 | 72 | 149
  Male | 20 | 27 | 47

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction In Systolic Blood Pressure (SBP) After 18 Weeks of Treatment From Baseline
Description: Baseline was defined as the latest SBP under monotherapy.
Time Frame: Baseline, Week 18
Population: MITT analysis set was defined as all randomized and treated subjects with at least 1 SBP measurement after the date of first dose of IMP. Here "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- Bisoprolol Failed Group: Subjects who failed monotherapy with bisoprolol 5 mg before trial inclusion were randomized to bisoprolol failed group to receive Bisoprolol/Amlodipine FDC tablet. Bisoprolol/Amlodipine FDC tablet was orally administered at an initial dose of 5 mg/5 mg once daily for 6 weeks. If BP was controlled at Week 6 (Day 43), the same dose was continued for next 6 weeks. If the BP was not controlled at Day 43, the dose was increased to Bisoprolol/Amlodipine 5 mg/10 mg or 10 mg/5 mg for next 6 weeks. Subjects who had controlled BP at Week 12 (Day 85), continued with the same dose that they were receiving for next 6 weeks. If their BP was not controlled at Day 85, dose was increased to the next level (Bisoprolol/Amlodipine 5 mg/10 mg for subjects receiving Bisoprolol/Amlodipine 5 mg/5 mg dose and Bisoprolol/Amlodipine and 10 mg/10 mg for subjects receiving Bisoprolol/Amlodipine 5 mg/10 mg dose) until Week 18 (Day 127). Controlled BP= SBP <140 mmHg and DBP <90 mmHg.
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group
Number analyzed (Participants) | 92 | 94
millimeters of mercury (mmHg)
  Baseline | 150.6 (8.21) | 151.6 (11.57)
  Change at Week 18 | -24.7 (11.67) | -25.9 (12.82)
Statistical Analysis 1: Comparison: Amlodipine Failed Group vs Bisoprolol Failed Group; For each group (Amlodipine failed and Bisoprolol failed) SBP after 18 weeks compared to baseline (under monotherapy). Superiority was assessed between FDC and monotherapies; Test type: Superiority or Other; p < 0.001, Paired t test — P value in both groups (Amlodipine failed and Bisoprolol failed) for comparison of SBP after 18 weeks versus baseline

2. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) After 18 Weeks of Treatment
Description: Baseline was defined as the latest DBP before study treatment administration.
Time Frame: Baseline, Week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group
Number analyzed (Participants) | 92 | 94
mmHg
  Baseline | 90.5 (6.92) | 92.0 (8.81)
  Change at Week 18 | -13.0 (9.38) | -14.0 (7.73)

3. Secondary Outcome: Percentage of Subjects With Controlled Blood Pressure
Time Frame: Baseline up to Week 18
Population: MITT analysis set included all randomized and treated subjects with at least 1 SBP measurement after the date of first dose of IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group
Number analyzed (Participants) | 97 | 99
percentage of subjects
  Week 6 | 85.6 | 80.8
  Week 12 | 86.8 | 87.9
  Week 18 | 86.7 | 89.0

4. Secondary Outcome: Change From Baseline in Heart Rate (HR) After 18 Weeks of Treatment
Description: Baseline was defined as the latest HR before study treatment administration
Time Frame: Baseline, Week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group
Number analyzed (Participants) | 89 | 94
beats per minute
  Baseline | 73.6 (8.96) | 69.9 (9.70)
  Change from baseline at Week 18 | -11.5 (8.65) | -6.6 (9.67)

5. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, AEs Leading to Discontinuation and AEs Leading to Death
Description: An AE was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent AEs was AEs that started or worsened in severity on or after the date of first dose of IMP until the end of the study. AEs leading to death and discontinued were also presented.
Time Frame: Baseline up to Day 127 (end of trial)
Population: Safety analysis set included all subjects who received at least 1 dose of IMP.
Measure: Number; unit: subjects
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group
Number analyzed (Participants) | 100 | 100
subjects
  TEAEs | 78 | 71
  Serious TEAEs | 1 | 2
  AEs leading to discontinuation | 3 | 3
  AEs leading to death | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 127
Arm/Group | Amlodipine Failed Group | Bisoprolol Failed Group
Serious Adverse Events (participants affected / at risk) | 1/100 | 2/100
Other Adverse Events (participants affected / at risk) | 63/100 | 53/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine Failed Group (N=100) | Bisoprolol Failed Group (N=100)
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine Failed Group (N=100) | Bisoprolol Failed Group (N=100)
Sinus bradycardia (Cardiac disorders) | 30 | 25
Bradycardia (Cardiac disorders) | 20 | 15
Oedema peripheral (General disorders) | 9 | 9
Urinary tract infection (Infections and infestations) | 6 | 9
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Overdose (Injury, poisoning and procedural complications) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No